CLINICAL TRIAL: NCT03535896
Title: Heavy-slow Resistance Training in Addition to an Ultrasound-guided Corticosteroid Injection to Reduce Pain in Individuals With Plantar Fasciopathy: a Feasibility Study
Brief Title: Heavy-slow Resistance Training and Ultrasound-guided Corticosteroid Injection in Plantar Fasciopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Henrik Riel, PhD student, Aalborg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018-521-0008
Record Dates: First submitted 2018-04-23; First posted 2018-05-24 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Plantar Heel Pain; Plantar Fasciopathy
MeSH Terms: interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HSR and injection (Experimental): HSR and corticosteroid injection
  Interventions: Other: HSR; Drug: Corticosteroid injection

INTERVENTIONS:
Other: HSR — Participants will complete a heel raise standing with the forefoot on a step. The toes are maximally dorsiflexed by placing a towel underneath them. The heel raise is performed with a raise to maximal plantar flexion and to maximal dorsi flexion.
  The exercise is performed with a load as heavy as possible but no heavier than 8RM and for as many sets as possible every other day.
Drug: Corticosteroid injection — Participants receive an ultrasound-guided corticosteroid injection between 5 and 8 days after baseline. A 21-gauge, 40 mm needle is connected to a 2.5 cm3 syringe filled with 1 ml Triamcinolonhexacetonid (Lederspan, Meda) + 1 ml Lidocain 10 mg7ml (Xylocain, AstraZeneca). The skin is cleansed with Chlorhexidine alcohol 0.5 % (Medic). The needle is inserted with a medial approach under ultrasound-guidance aligned to the long axis of the ultrasound transducer. The injection is placed anterior to the plantar fascia insertion on the calcaneal bone in the region of maximal fascia thickness.

SUMMARY:
The purpose of this study is to investigate the feasibility of combining heavy-slow resistance training with an ultrasound-guided corticosteroid injection to reduce pain in individuals with plantar fasciopathy. Feasibility will be evaluated using the acceptability of the combined interventions and exercise compliance.

DETAILED DESCRIPTION:
After eligibility has been confirmed, participants are instructed in performing the exercise which will be heel raises. Participants will be asked to complete the exercise standing with the forefoot on a step. The toes are maximally extended by placing a towel underneath them. The participant is instructed to perform a heel raise to maximal plantar flexion in the ankle joint and afterwards to lower the heel to maximal dorsiflexion. Supporting oneself for balance by touching the hands on a wall or a rail is allowed. The participants are instructed in performing the exercise with a load as heavy as possible but no higher than 8RM and for as many sets as possible. If the participants feel they can perform more repetitions than their load corresponds to (e.g. 10 repetitions when the load is supposed to be 8RM) an external load consisting of a backpack with books or water bottles to add weight will be used. Participants are asked to start performing the exercise as soon as they feel ready but not before 24 hours after the injection.

Participants will receive patient education on what is known about the condition in terms of risk factors and aetiology, the pathology, activity modification, and the rationale for why the combination of heavy slow resistance training and an US-guided corticosteroid injection could lead to recovery. They will be told that compliance to the exercise programme is very important and that compliance to the exercises is associated with their recovery. They are also informed about other types of evidence-based treatments however, they are asked to refrain from seeking other treatments during the course of the study. A silicone heel cup will be given to all participants and they are asked to use the heel cup as much as possible. If the participant already uses an insole or any other type of foot orthosis they will be allowed to continue wearing this if they do not want to use the heel cup. Participants are asked not to progress the method used to achieve 8RM when they start to do the exercise after the injection until Week 3 of the exercise program. If standing on both feet was sufficient to achieve 8RM at baseline, the participant must not perform the exercise single-legged after the injection regardless of any pain reduction afforded by the injection.

Participants receive an ultrasound-guided corticosteroid injection between 5 and 8 days after baseline. A 21-gauge, 40 mm needle is connected to a 2.5 cm3 syringe filled with 1 ml Triamcinolonhexacetonid (Lederspan, Meda) + 1 ml Lidocain 10 mg7ml (Xylocain, AstraZeneca). The skin is cleansed with Chlorhexidine alcohol 0.5 % (Medic). The needle is inserted with a medial approach under ultrasound-guidance aligned to the long axis of the ultrasound transducer. The injection is placed anterior to the plantar fascia insertion on the calcaneal bone in the region of maximal fascia thickness. If participants are not categorised as improved based on the Global Rating of Change after the 8 weeks of exercise they will be offered to receive a second injection and are advised to continue performing the exercise. These participants will have an additional follow-up 8 weeks after the second injection.

All statistical analyses will be performed according to a pre-established analysis plan. STATA ver. 14 will be used as statistical software.

Feasibility outcomes To conclude that the combined interventions are feasible the following three criteria will need to be met: i) ≥10/20 rate the combined interventions as "acceptable". The rationale for choosing this criterion is that the effect of the combined interventions has yet to be established and effective treatment could justify the use of an intervention that is slightly uncomfortable or considered slightly unacceptable by patients (e.g. chemo therapy is a very uncomfortable treatment but is tolerated and accepted by patients because of the potential effective outcome). Any dropouts after the injection will be dichotomized as "unacceptable". ii) based on the self-reported training diaries ≥15/20 participants will need to have performed ≥20/27 possible training sessions; and iii) ≥15/20 participants will need to have started performing the exercise ≤7 days after the injection. Weekly recruitment rate will be reported using descriptive statistics.

Explorative quantitative outcomes Any changes in FHSQ, IPAQ, and PSEQ will be examined using a one-way repeated measures ANOVA, with time (baseline assessment, 4 weeks, or 8 weeks) as the independent factor, and FHSQ, IPAQ or PSEQ, respectively, as the dependent variable. Changes in plantar fascia thickness from baseline assessment to the 8-week follow-up and the difference in mean daily heel pain from before to after the injection will be examined using paired t-tests. GROC will be reported using descriptive statistics.

If any participant decides to drop out before having received the injection a new participant will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* History of inferior heel pain for at least three months before enrolment
* Pain on palpation of the medial calcaneal tubercle or the proximal plantar fascia
* Thickness of the plantar fascia of 4 mm or greater
* Mean heel pain of 30 mm or above on a 0 to 100 mm VAS during the previous week

Exclusion Criteria:

* Below 18 years of age
* History of inflammatory systemic diseases
* Prior heel surgery
* Pregnancy
* Pain or stiffness in the 1st metatarsophalangeal joint to an extent where the exercises cannot be performed
* Corticosteroid injection for plantar fasciopathy within the previous six months
* Known hypersensitivity to corticosteroids or local anaesthetics
* Skin or soft tissue infection near the injection site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2018-10-11 (Actual)

PRIMARY OUTCOMES:
Acceptability | At the 8-week follow-up
  Acceptability of the combined interventions measured by a participant acceptability questionnaire that includes a 7-point Likert scale ranging from "very unacceptable" to "very acceptable". This is not a measure of whether the participant's symptoms have improved to a point where they are recovered or feel close to recovery but if it matches their expectations to the content of the intervention and acceptability of performing exercise after receiving an injection. This will be clearly stated on the questionnaire to emphasise that improvement is not to be considered. The combined interventions are categorised as "unacceptable" if they are rated as "very unacceptable" or "unacceptable" (category 1-2) and categorised as "acceptable" if they are rated from "slightly unacceptable" to "very acceptable" (category 3-7).
Compliance | From baseline to the 8-week follow-up
  Compliance to the exercises as measured by the mean number of training sessions performed per week throughout the intervention measured by a training diary that each participant is handed out at baseline. The participants will be instructed in filling out the number of repetitions and sets performed and the day on which they performed the exercise
Recruitment rate | From start of recruitment until the 20th participant has been recruited, assessed up to 12 months
  Mean number of participants recruited per week
Exercise start | From date of injection to exercise start assessed up to 8 weeks
  Mean days until the participant starts to perform the exercises from the two days after the injection based on training diary data. Participants are asked to start performing the exercise as soon as they feel ready but not before two days after the injection.

SECONDARY OUTCOMES:
Change in Foot Health Status Questionnaire | At baseline and at the 4- and 8-week follow-ups
  Ranging from 0 (poor foot health) to 100 (optimum foot health)
Change in mean daily heel pain measured on an 11-point Numerical Rating Scale (NRS) | From baseline to one week after injection
  Participants receive a daily SMS asking them to rate their mean heel pain during the past 24 hours on an NRS (ranging from 0 (no pain) to 10 (worst pain imaginable)) from the day after baseline to one week after the injection
Global Rating of Change | At the 8-week follow-up
  This will be used to measure the participants' self-reported recovery on a 7-point Likert scale ranging from "much improved" to "much worse". Participants are categorised as improved if they rate themselves as "much improved" or "improved" (category 6-7) and categorised as not improved if they rate themselves from "slightly improved" to "much worse" (category 1-5).
Change in plantar fascia thickness | At baseline and at the 8-week follow-up
  Measured in millimeters using ultrasonography
Change in Pain Self-Efficacy Questionnaire score | At baseline and at the 4- and 8-week follow-ups
  The Pain Self-Efficacy Questionnaire ranges from 0 (not at all confident) to 60 (completely confident) with lower scores indicating lower self-efficacy. A Danish translation of the original questionnaire, which has been validated in a Danish chronic pain population, will be used.
Change in physical activity level | At baseline and at the 4- and 8-week follow-ups
  This will be measured using the International Physical Activity Questionnaire short form (IPAQ). A Danish translation of the original questionnaire will be used. The IPAQ is the most commonly used questionnaire for measuring physical activity among adults and consists of 9 items that provide information on the time spent performing vigorous and moderate activities, the time spent walking, and time spent sedentary during the past week. The IPAQ gives an estimate of the total weekly physical activity measured in MET-minutes per week and total minutes spent sitting

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Riel, MSc, Principal Investigator — Research Unit for General Practice in Aalborg, Department of Clinical Medicine, Aalborg University
Locations (1):
- Research Unit for General Practice in Aalborg, Department of Clinical Medicine, Aalborg University, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Riel H, Olesen JL, Jensen MB, Vicenzino B, Rathleff MS. Heavy-slow resistance training in addition to an ultrasound-guided corticosteroid injection for individuals with plantar fasciopathy: a feasibility study. Pilot Feasibility Stud. 2019 Aug 24;5:105. doi: 10.1186/s40814-019-0489-3. eCollection 2019. PMID 31463078